CLINICAL TRIAL: NCT06344598
Title: Clinical and Epidemiological Risk Evaluation of Osteoporosis Prevalence at Different Ages With to Assess Bone Quantification Using Dual-energy X-ray Absorptiometry
Brief Title: Identification and Assessment of Risk Factors for the Development of Osteoporosis in Adults and Children Living in the Abay Region of the Republic of Kazakhstan Using the Method of Dual-energy X-ray Absorptiometry and Clinical and Epidemiological Research
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semey State Medical University (Other)
Collaborators: Ministry of Science and Higher Education of the Republic of Kazakhstan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0123РК00314; AP19680262 (Other: Science Committee of the Ministry of Science and Higher Education of the Republic of Kazakhstan)
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-09

CONDITIONS: Improving the Early Diagnosis of Osteoporosis in Adults and Children Living in the Abay Region of Kazakhstan
Keywords: osteoporosis, dual-energy X-ray absorptiometry, bone mineral density, risk factors
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persons with normal BMD
- Persons with low BMD

SUMMARY:
A survey of people to identify risk factors for osteoporosis, which include age, gender, lifestyle, diet, physical activity, the presence or absence of somatic pathology. Diagnosis of osteoporosis by dual-energy X-ray absorptiometry. Conducting a correlation analysis of the relationship of the data obtained.

DETAILED DESCRIPTION:
Successful diagnosis of osteoporosis is possible with the complex use of clinical, laboratory and radiological methods. In the complex of diagnostic methods, a special place has given to dual-energy X-ray absorptiometry, which is the "gold standard". The research area contains the following tasks:

Risk factors for the development of osteoporosis will be identified and quantified in the formed study groups of adults; to determine the diagnostic value of the risk factors for the development of osteoporosis obtained during the examination.

to assess the state of BMD in adults using X-ray absorptiometry (DXA) To carry out a correlation analysis of the relationship between the obtained data in adults of the Abay region of of the Republic of Kazakhstan

ELIGIBILITY:
Inclusion Criteria: adults and children without a history of pathological fractures and congenital pathology of the musculoskeletal system.

-

Exclusion Criteria: adults and children with congenital pathology of the musculoskeletal system

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of the Abay region of the Republic of Kazakhstan
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk factors for the development of osteoporosis will be identified and quantified in the formed study groups of adults | By the end of Dec 2025
to determine the diagnostic value of the risk factors for the development of osteoporosis obtained during the examination | By the end of Dec 2025
to assess the state of BMD in adults using X-ray absorptiometry (DXA) | By the end of Dec 2025
To carry out a correlation analysis of the relationship between the obtained data in adults of the Abay region of of the Republic of Kazakhstan | By the end of Dec 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Semey Medical University, Semey, Kazakhstan